CLINICAL TRIAL: NCT05099588
Title: The Incidence of Treatment-requiring Retinopathy of Prematurity in Greece: a Multicenter Prospective Cohort Study
Brief Title: The Incidence of Treatment-requiring Retinopathy of Prematurity in Greece
Acronym: GR-ROP
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Athens General Children's Hospital "Pan.&Aglaia Kyriakou", Athens, Greece (Unknown); Agia Sofia Children's Hospital, Athens, Greece (Unknown); Attikon Hospital (Other); Iaso Neonatology Clinic, Athens, Greece (Unknown); REA Maternity Hospital, Athens, Greece (Unknown); Ippokratio General Hospital, Thessaloniki, Greece (Unknown); General University Hospital of Patras, Greece (Unknown); General University Hospital of Larisa, Greece (Unknown); University Hospital, Ioannina (Other); General University Hospital of Heraklion, Greece (Unknown); Venizeleio General Hospital of Heraklion, Greece (Unknown); General University Hospital of Alexandroupoli, Greece (Unknown)
Responsible Party: Principal Investigator, Asimina Mataftsi, Associate Professor in Ophthalmology, Paediatric Ophthalmology and Strabismus, Aristotle University Of Thessaloniki
Other Study IDs: 280/15-04-2020
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of prematurity; ROP; Treatment
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants treated for ROP
  Interventions: Other: Other: observational study

INTERVENTIONS:
Other: Other: observational study — Observational study

SUMMARY:
A prospective observational study of the incidence of treatment-requiring ROP (TR-ROP), at a national level, in Greece.

DETAILED DESCRIPTION:
The purpose of this observational study is to prospectively collect data on ROP cases necessitating treatment at a national level. Each and every ROP screening unit in Greece (collaborating centers) report their new TR-ROP cases, their demographics and treatment characteristics, monthly, for a 12-month period. A reminder email is sent to avoid under-reporting due to neglect. Data are collected by the Responsible Party and will be analyzed together with national registry data on all preterm births in the same 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants undergoing screening for ROP, who developed TR-ROP and were treated for ROP in one or two eyes.

Exclusion Criteria:

* None.

Ages: 30 Weeks to 50 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants who underwent treatment for ROP in a public or private hospital in Greece during the 12-month study period.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-requiring ROP (TR-ROP) in Greece | During the study period (1 year, prospectively)

SECONDARY OUTCOMES:
The mean gestational age and birth weight of infants treated for ROP in Greece | During the study period (1 year, prospectively)
The rate of participants treated with laser photocoagulation versus anti-VEGF injection | During the study period (1 year, prospectively)
The failure and recurrence rate of applied treatments for ROP | During the follow-up period (6 months from treatment, prospectively)

CONTACTS AND LOCATIONS:
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams GG, Bunce C, Xing W, Butler L, Long V, Reddy A, Dahlmann-Noor AH. Treatment trends for retinopathy of prematurity in the UK: active surveillance study of infants at risk. BMJ Open. 2017 Mar 21;7(3):e013366. doi: 10.1136/bmjopen-2016-013366. PMID 28325857